CLINICAL TRIAL: NCT05081505
Title: The Influence of a New Intervention Model of Community-based Physical Fitness Exercise on the Older Adults' Adherence to Physical Activity and the Improvement of Functional Fitness
Brief Title: Community-based Physical Fitness Exercise on the Older Adults' Functional Fitness and Adherence to Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KMUHIRB-E(II)-20190397
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Older Adult

STUDY DESIGN:
Intervention Model Description: This is a single group trial, according to the pre-test result of the exercise stage of the change questionnaire, they were divided into the maintenance phase group (MP, N=15) and under the maintenance phase group (MPb, N=15). All subjects joined the community-based physical fitness exercise course for 24 weeks. To quantify the effect of this intervention method on functional fitness and exercise persistence of the elderly, this study analyzed the related exercise behavior changes of MPb and MP elderly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-based physical fitness exercise course (Experimental): Included 12-week structural exercise course (0-12 weeks) and 12-week autonomous group class (12-24 weeks).
  Interventions: Behavioral: Structural exercise course; Behavioral: Autonomous group class

INTERVENTIONS:
Behavioral: Structural exercise course — 12-week structured exercise class, team competition, social support, and incentive strategy
Behavioral: Autonomous group class — 12-week autonomous group class, team competition, social support, and incentive strategy

SUMMARY:
Maintaining adequate physical activity (PA) and regularly exercising are very important to promote the good physical and mental health of the elderly. According to the transtheoretical model (TTM) framework, previous research studies have formulated many strategies to promote exercise behaviors, such as incentive strategies, combines municipal resources and links up with the referral of primary care institutions, or including patients in the decision-making process about exercise choices to enable patients to have greater autonomy. In addition, in terms of the strategic aspects of achieving goals, competitive incentives are also an effective strategy. Therefore, this study aims to find out the effects of the community-based physical fitness exercise course, which is given according to TTM, on improving functional fitness and exercise persistence of the older adults.

ELIGIBILITY:
Inclusion Criteria:

* age between 65 to 90 years old
* can stand up from a chair without armrests
* can walk independently for 2 minutes without relying on any mechanical assistance
* no medical issues according to the PAR-Q+ form assessment
* can complete the Senior Fitness Test (SFT)

Exclusion Criteria:

* diagnosed with severe dementia (unable to understand and/or follow verbal commands)
* suffering from stroke, severe hypertension, heart disease, and diabetes
* hip or knee replacement surgery in the past 6 months
* hip fracture
* having undergoing rehabilitation plan
* unable to complete the pre-tests or post-test

Ages: 65 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Exercise stage of change questionnaire | basal, 12, 24 weeks follow up
  Exercise Change Stage Short Question Form is a 5 item scale. It has only one question, used to categorizes individuals into one of the five stages of change: (1) Precontemplation (2) Contemplation (3) Preparation (4) Action (5) Maintenance.
Physical Activity Scale for the Elderly (PASE) | basal, 12, 24 weeks follow up
  PASE is used to assess the physical activity level of elderly individuals, the factors affecting the activity level, the relationship between physical activity and health profile. The minimum and maximum score that can be obtained from the scale is 0 and 400.The higher score indicates better level of physical activity.
Exercise Self-efficacy Scale | basal, 12, 24 weeks follow up
  The Exercise Self-efficacy Scale measures an individual's perceived ability to overcome various obstacles to perform physical activity, with higher scores indicating more confidence in performing the exercise.
Outcome Expectations for Exercise Scale | basal, 12, 24 weeks follow up
  The Outcome Expectations for Exercise Scale contains 9 statements rated by participants using a 5-point Likert scale from 1 "Strongly Disagree" to 5 "Strongly Agree". It can help identify older adults with low outcome expectations for exercise.
Physical Activity Survey | basal, 12, 24 weeks follow up
  The physical activity survey is measured according to the PASE items. It is calculated by the frequency value (hours per day in the one-week reporting period) for low-intensity, medium-intensity, high-intensity, and muscle strengthening exercise. The higher score indicates the more time spent on the physical activity at each level.
Attendance rate | 12 and 24 weeks
  The attendance rate of the subjects participating in structured exercise courses and autonomous group classes
Senior Fitness Test - Body Mass Index (BMI) | basal, 12, 24 weeks follow up
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Senior Fitness Test - Waist-hip ratio | basal, 12, 24 weeks follow up
  The waist-hip ratio is the dimensionless ratio of the circumference of the waist to that of the hips.
Senior Fitness Test - 30s Chair stand | basal, 12, 24 weeks follow up
  Evaluates the lower body strength according to the number of times the individual stood up and sat down in 30 seconds. Characterized as continuous numeric variable
Senior Fitness Test - Chair Sit-&-Reach | basal, 12, 24 weeks follow up
  Evaluates the lower back and hamstring flexibility according to the distance measured between the tip of the finger tips and the toes. Characterized as continuous numerical variable.
Senior Fitness Test - 8-Foot Up-&-Go | basal, 12, 24 weeks follow up
  Assesses motor agility and dynamic balance. Evaluates the time in seconds and hundredths in an established path of 2.44 meters on the route to go and return to starting position. Characterized as continuous numerical variable.
Senior Fitness Test - 30s Arm curl | basal, 12, 24 weeks follow up
  Evaluates the upper body strength and endurance according to the number of arm curls in 30 seconds. Characterized as continuous numeric variable.
Senior Fitness Test - Back scratch | basal, 12, 24 weeks follow up
  Evaluates the flexibility of the upper limbs. It measures the distance in inches between the tips of the fingers in the back area. Characterized as continuous numeric variable
Senior Fitness Test - 2-Minute Step | basal, 12, 24 weeks follow up
  Evaluates aerobic endurance. Total double past stationary in 2 minutes. Characterized as continuous numeric variable.
Open-eyes one leg stand | basal, 12, 24 weeks follow up
  Evaluates the balance ability. The standing time on one leg, keep eyes open. Characterized as continuous numeric variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan